CLINICAL TRIAL: NCT03907735
Title: Oxytocin Receptor Expression in Pregnancy: When Does it Turn on
Brief Title: Oxytocin Receptor Expression in Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Reid, Instructor, Oregon Health and Science University
Other Study IDs: OHSU IRB 19417
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Post-Abortion; Hemorrhage, Obstetric
Keywords: Post-abortion hemorrhage; Obstetric hemorrhage; Preterm labor; Abnormal labor; Oxytocin; Oxytocin receptor
MeSH Terms: conditions — Hemorrhage; Obstetric Labor, Premature; Dystocia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Uterine biopsy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- 2nd trimester: Second trimester myometrial tissue samples will be collected by core needle biopsy under ultrasound guidance in anesthetized women. Samples will be obtained primarily after second trimester surgical abortions or Dilation and Evacuation (D&E) procedures as well as after rare gravid hysterectomies or after late second trimester cesarean deliveries.
  Interventions: Other: Myometrial tissue sample collection
- Non-pregnant: Myometrial tissue samples will be collected by core needle biopsy under ultrasound guidance in non-pregnant women undergoing gynecologic surgery under anesthesia for laparoscopic tubal ligation.
  Interventions: Other: Myometrial tissue sample collection
- 1st trimester: First trimester myometrial tissue samples will be collected by core needle biopsy under ultrasound guidance in anesthetized women. Samples will be obtained after first trimester surgical abortions or suction dilation and curettage (D&C).
  Interventions: Other: Myometrial tissue sample collection
- After term pregnancy (3rd trimester): Third trimester myometrial tissue samples will be collected by core needle biopsy under ultrasound guidance in anesthetized women. Samples will be obtained at the time of cesarean delivery.
  Interventions: Other: Myometrial tissue sample collection

INTERVENTIONS:
Other: Myometrial tissue sample collection — Myometrial tissue samples by core needle biopsy under ultrasound guidance

SUMMARY:
This study aims to determine when during gestation oxytocin receptor (OXTR) expression increases in the myometrium, which will contribute new insight to the management of obstetric hemorrhage and our understanding of normal and abnormal labor.

DETAILED DESCRIPTION:
In this descriptive study, we will obtain myometrial tissue samples by core needle biopsy under ultrasound guidance in anesthetized women immediately following surgical abortion and from controls, all of whom are undergoing a separate planned obstetric/gynecologic surgery. Tissue studies will be performed on these biopsy samples to examine oxytocin receptor expression and function.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-50
* Gestational age 14-26 weeks; or 6-13 weeks, 37-42 weeks, or non-pregnant (controls)
* Undergoing another planned surgical procedure with anesthesia (suction D&C, D&E, gravid hysterectomy, cesarean section, or laparoscopic tubal ligation)
* Able to give informed consent in English or Spanish

Exclusion Criteria:

To optimize biopsy safety, we will exclude patients with anticipated difficult cases, that have additional risks of hemorrhage, or those with features that limit ultrasound visualization.

Increased risk of hemorrhage:

* Anemia (Hgb < 9)
* Anticoagulation, bleeding disorder, or coagulopathy
* Multiple gestation
* Infection or sepsis

For ultrasound-guided procedures:

* Obese, BMI ≥ 40
* History of ≥2 cesarean sections
* Large fibroids or uterine anomalies obstructing view
* Other poor visualization
* Thin myometrium < 1cm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a study of reproductive age women over 18 years of age being performed at Oregon Health & Science University (OHSU) in Portland, OR. It will include subjects who present for pre-operative appointments in our outpatient Center for Women's Health Family Planning Clinic and OHSU Labor and Delivery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Oxytocin receptor expression | 30 minutes
  Measure of oxytocin receptor expression. Perform quantitative RT-PCR on mRNA extracted from biopsy samples obtained from subjects at the end of their procedure (within 30 minutes).

SECONDARY OUTCOMES:
Function of myometrial oxytocin receptor | 30 minutes
  Assessment of the function of the myometrial oxytocin receptor. Measure intracellular calcium in cultured myometrial cells after activating the receptor with oxytocin from biopsy samples obtained from subjects at the end of their procedure (within 30 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Reid, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No